CLINICAL TRIAL: NCT03618667
Title: A Phase II Clinical Study of GC1118 in Recurrent Glioblastoma Patients With High Epidermal Growth Factor Receptor (EGFR) Amplification
Brief Title: GC1118 in Recurrent Glioblastoma Patients With High EGFR Amplification
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Se-Hoon Lee, Professor, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMC2017-06-111
Record Dates: First submitted 2018-07-07; First posted 2018-08-07 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2022-11

CONDITIONS: Glioblastoma, Adult; EGFR Amplification
MeSH Terms: conditions — Glioblastoma | interventions — GC1118

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single group (Experimental): GC1118 (4mg/kg) will be administered by IV infusion once per week for 4 weeks(28-day cycle) up to 6 cycles, or till progression or uncontrolled toxicity.
  Interventions: Drug: GC1118

INTERVENTIONS:
Drug: GC1118 — GC1118 (4mg/kg) will be administered by IV infusion once per week for 4 weeks(28-day cycles) up to 6 cycles, or till progression or uncontrolled toxicity.

SUMMARY:
This study is a phase 2 trial of GC1118, an EGFR monoclonal antibody, for recurrent glioblastoma patients who were treated with standard concurrent chemoradiation.

DETAILED DESCRIPTION:
This study is a phase 2 trial of GC1118, an EGFR monoclonal antibody, for recurrent glioblastoma patients who were treated with standard concurrent chemoradiation.

GC1118 (4mg/kg) will be administered by IV infusion once per week for 4 weeks(28-day cycle) up to 6 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. written informed consent
2. 19 years or older
3. patients who experience recurrence following the standard therapy (CCRT, adjuvant temozolomide)
4. high EGFR amplification
5. available archive tumor sample(s)
6. Karnofsky performance status (KPS) > 70
7. life expectancy > 3 months
8. adequate end-organ function
9. patients who recovered from previous therapy (NCI CTCAE v4.03 Gr 1)

Exclusion Criteria:

1. patients who had EGFR target agent(s) before screening
2. patients who have clinically significant cardiopulmonary dysfunction (cardiovascular disease (> 2grade, NYHA), myocardial infarction within previous 3 months, unstable angina, unstable arrythmia, clinically significant interstitial lung disease)
3. patients who had major surgery, open biopsy, or clinically significant trauma within previous 4 weeks
4. patients who had investigation drug(s) within previous 4 weeks
5. patients who had other malignancy(ies) within previous 3 years (except malignancies with low tendency to metastases or mortality for example, treated cervical intraepithelial neoplasia, skin cancer except melanoma, localized prostate cancer)
6. patients who had severe infection within previous 4 weeks
7. HIV infection
8. patients who had anti-cancer therapy (surgery, chemo-radiation, chemotherapy, radiation therapy) within previous 4 weeks
9. clinically significant liver disease (active hepatitis B viral (HBV) or hepatitis C viral (HCV) infection, alcoholic liver disease etc)
10. pregnancy or breast-feeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2018-09-08 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | at 6 months
  survival time from screening to progression defined by RANO criteria

SECONDARY OUTCOMES:
overall survival | 6 months, 12 month
  survival time from screening to death of any cause
overall response rate | up to 30months
  best overall response rate defined by RANO criteria
Exploration of predictive/prognostic biomarkers | up to 30 months
  according to NGS-based biomarkers(whole exome sequencing and whole transcriptome sequencing)

CONTACTS AND LOCATIONS:
Overall Officials: sehoon lee, professor, Study Director — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided